CLINICAL TRIAL: NCT05875857
Title: Patient Utilization of Opioid Destruction Bags in the Post-op Period
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0277-22-EP
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use; Opioid Use, Unspecified; Patient Empowerment; Total Knee Arthoplasty; Total Hip Arthroplasty
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group will receive current standard of care education and surveys at 6-8 weeks post discharge.
- Intervention (Experimental): Intervention group will receive a specialized handout and patient education on the safe storage of opioid medications, importance of opioid destruction, opioid destruction options and medication destruction (Deterra) bag before discharge. Surveys will be sent to group at 6-8 weeks post discharge.
  Interventions: Behavioral: Opioid destruction education

INTERVENTIONS:
Behavioral: Opioid destruction education — Intervention group will receive a specialized handout and patient education on the safe storage of opioid medications, importance of opioid destruction, opioid destruction options and medication destruction (Deterra) bag before discharge.
  Arms: Intervention

SUMMARY:
This is a study on how patients use and store opioid pain medications at home after surgery and what happens to left over pills when patients are done taking them. Participants will be taught the proper storage and destruction of opioid pain medications, then contacted in 6-8 weeks about pain medication used, stored disposed of.

DETAILED DESCRIPTION:
This is a randomized single-center prospective survey study to describe the utilization of opioid destruction bags in the post-operative period. Participants who underwent surgery for Total Knee Arthroplasty (TKA) or Total Hip Arthroplasty (THA) will be eligible for inclusion if discharging to home with an opioid prescription. Eligible participants will be randomized between two groups: 1) Control group will receive current standard of care 2) Intervention group will receive a specialized handout and patient education on the safe storage of opioid medications, importance of opioid destruction, opioid destruction options and medication destruction (Deterra) bag before discharge. Participants will be phoned/emailed six to eight weeks post-surgery to complete a survey. Attempts will be made on three separate days to reach the participant via phone. If email is preferred, three reminders will be sent to complete the survey. If participant is unreachable, they will be considered lost to follow up. Survey questions will be comprised of various question styles, including: yes/no, multiple choice, and free text answers.

ELIGIBILITY:
Inclusion Criteria:

19 years of age or older Discharging to home and prescribed opioids at discharge post total knee arthroplasty or total hip arthroplasty

Exclusion Criteria:

Under 19 years of age Opioid medication use prior to surgery Not prescribed an opioid to take after discharge

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Opioid destruction | Six to Eight weeks post discharge
  Number of patients who report they did or plan to destroy unused opioids

SECONDARY OUTCOMES:
Patient Education | Six to Eight weeks post discharge
  Number of patients who recall patient education on storage and disposal of opioid medications at discharge
Opioid Storage | Six to Eight weeks post discharge
  Type of opioid storage method used at home
Opioid Destruction Method | Six to Eight weeks post discharge
  Type of opioid destruction method used or plan to use
Leftover Pills | Six to Eight weeks post discharge
  Estimated number of pills leftover after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kristin R Daniel, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No